CLINICAL TRIAL: NCT04012099
Title: An Independent Evaluator-Blind, Dose-Escalation, Untreated-Controlled, Within-Subject, Phase 2a Therapeutic Exploratory Clinical Trial to Evaluate the Efficacy and Safety of BMT 101 Administration for the Prevention of Hypertrophic Scar
Brief Title: the Hypertrophic Scar Prevention of BMT101.
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Internal reasons
Sponsor: Hugel (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Prevention
Other Study IDs: HG-BMT-PIIa-01
Record Dates: First submitted 2018-12-03; First posted 2019-07-09 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2022-07

CONDITIONS: Hypertrophic Scar
Keywords: scar prevention; siRNA; scar
MeSH Terms: conditions — Cicatrix, Hypertrophic; Cicatrix

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BMT101 (Experimental): BMT101 injection (treatment)
  Interventions: Drug: BMT101
- control (No Intervention): Un-treated control

INTERVENTIONS:
Drug: BMT101 — Intradermal injection to each of 3 dose-groups.
  Other Names: cp-asiRNA
  Arms: BMT101

SUMMARY:
An Independent Evaluator-Blind, Dose-Escalation, Untreated-Controlled, Within-Subject, Phase 2a Therapeutic Exploratory Clinical Trial

DETAILED DESCRIPTION:
As a comparative evaluation between the control group (untreated-control) and the study group (treatment) within a subject, it was decided to assign ten subjects to each of the three dose groups.

ELIGIBILITY:
Inclusion Criteria:

* male and female adults aged 19-55 years
* Those who plan to undergo a revision surgery to remove hypertrophic scar resulted from a previous abdominal surgery
* Those who voluntarily signed the written consent and agreed to participate in the study.

Exclusion Criteria:

* Pregnant or lactating women
* Those with clinically significant systemic disease (e.g. diabetes, hematologic disease, allergic or immunogenic systemic skin disease)

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2019-08-21 (Actual); Primary Completion 2023-05-10 (Actual); Study Completion 2023-05-10 (Actual)

PRIMARY OUTCOMES:
Reducing the hypertrophic scar after scar revision surgery | Week 2, 6, 10, 22
  to evaluate Differences in Visual Analogue Scale (VAS) score between the study group and the control group when independent evaluators assessed the severity of the hypertrophic scars.
Safety evaluation of BMT101 | Week 2, 6, 10, 22
  To assess severity and frequency of reported adverse events and clinically-relevant changes in laboratory testing after elective revision of a hypertrophic scar

CONTACTS AND LOCATIONS:
Locations (1):
- Hugel, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No